CLINICAL TRIAL: NCT00921245
Title: First REal-life Evaluation of Darifenacin in Overactive Bladder Patients During 3 Months
Brief Title: FREEDOM - First Real-Life Evaluation of Enablex Done in ZA Overactive Bladder Patients During a 3 Months Period
Acronym: FREEDOM
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Healthcare AG
Other Study IDs: 13027; EX0710ZA (Other: Company internal)
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — darifenacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Darifenacin (Emselex, BAY79-4998)

INTERVENTIONS:
Drug: Darifenacin (Emselex, BAY79-4998) — Patients in daily clinical treatment receiving Emselex according to local drug information

SUMMARY:
Patient perspective on Overactive Bladder and symptoms experienced after administration of Darifenacin

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients > 18 years with symptoms of overactive bladder.

Exclusion Criteria:

* Contraindications for the treatment with Darifenacin prolonged-release tablets according to the registered package insert.
* Pregnancy and lactation. Women of childbearing potential have to use an acceptable method of contraception.
* Concomitant treatment with drugs known to affect mainly the urinary bladder function (e.g. anticholinergics, antispasmodics) at any time during the study. Concomitant treatment with botulinum toxin, capsaicin or resiniferatoxin at any time during the study and treatment with botulinum toxin, capsaicin or resiniferatoxin in the last 6 months prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Private Practice Patients
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of Darifenacin in the daily practice for the treatment of the OAB (Over Active Bladder) syndrome. | 3 months later

SECONDARY OUTCOMES:
To evaluate the patient's perception of bladder condition, the patient's use of the patient support program, the patient's and physician's assessment of treatment regarding efficacy and tolerability and patient's compliance with the treatment | 3 months later

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Africa